CLINICAL TRIAL: NCT06082141
Title: Contribution of Transversus Thoracis Plane Block in Combination With Serratus Anterior Plane Block to the Quality of Recovery After Breast Cancer Surgery: a Randomized Controlled Trial
Brief Title: Effect of Adding TTPB to SAPB in Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Aylin Ceren Sanli, Asist Dr, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E.116140
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain; Opioid Use
Keywords: Quality of recovery-15; Serratus anterior plan block; Transversus thoracis plan block
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided serratus anterior plane block (Active Comparator): SAP block will be made with 10 ml 0.5% bupivacaine + 10 ml NaCl TTP block will be made with 10 ml NaCl
  Interventions: Procedure: Serratus anterior plan block
- Combination of ultrasound-guided serratus anterior plane block and transversus thoracis plane block (Active Comparator): SAP block will be made with 10 ml 0.5% bupivacaine + 10 ml NaCl TTP block will be made with 5 ml 0.5% bupivacaine + 5 ml NaCl
  Interventions: Procedure: Transversus thoracis plane block combined with serratus anterior plane block

INTERVENTIONS:
Procedure: Transversus thoracis plane block combined with serratus anterior plane block — SAP block will be made with 10 ml 0.5% bupivacaine + 10 ml NaCl under US-guidance, TTP block will be made with 5 ml 0.5% bupivacaine + 5 ml NaCl under US-guidance
  Arms: Combination of ultrasound-guided serratus anterior plane block and transversus thoracis plane block
Procedure: Serratus anterior plan block — SAP block will be made with 10 ml 0.5% bupivacaine + 10 ml NaCl under US-guidance, TTP block will be made with 10 ml NaCl under US-guidance
  Arms: Ultrasound guided serratus anterior plane block

SUMMARY:
Breast cancer is the most common malignancy in women worldwide. Even minor breast surgery can cause significant postoperative pain (PP). PP can turn into chronic pain in 25-40% of cases. Inadequate PP control is associated with increased morbidity, delayed wound healing, prolonged hospital stay, increased opioid use and side effects, and high cost of care.

Opioid use remains the mainstay of postoperative analgesia. Opioids, especially morphine, inhibit both cellular and humoral immune functions. This effect may be responsible for the high rates of local recurrence and/or metastasis after surgery. Additionally, studies have shown that perioperative opioid use is associated with social abuse. This demonstrates the importance of reducing perioperative opioid use. Currently, multimodal analgesia based on nerve block is being widely investigated and has shown encouraging clinical results.

Numerous regional analgesic techniques have been investigated in breast cancer surgery, including intercostal nerve block, thoracic epidural anesthesia, and paravertebral block. Compared with general anesthesia alone, it reduces the postoperative pain score even after a single-shot injection for up to 72 hours, reduces opioid consumption, improves the quality of patient recovery, and suppresses the development or reduces the severity of chronic pain.

Serratus anterior plane block (SAPB) is reported to be effective in perioperative pain management of breast cancer surgeries. The important problem of SAPB block is that it is insufficient to block the anterior cutaneous branches of the intercostal nerves. Therefore, intravenous analgesia is required. Thoracic transversus muscle plane block (TTPB) is a recently described fascial plane block used to anesthetize the anterior cutaneous branches of the intercostal nerves from T2-T6. Its effectiveness has been demonstrated for breast surgery and median sternotomy.

In our study, we will provide postoperative analgesia in patients undergoing breast surgery by applying the serratus anterior block in combination with the transversus thoracis plane block. Since we avoid complicated analgesia methods such as paravertebral block, the risk of complications will be reduced.

In this study, we aimed to compare the effectiveness of the combination of SAPB and TTPB with SAPB performed alone in breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* BMI 20 to 35 kg / m2
* Patients scheduled for breast cancer surgery procedure

Exclusion Criteria:

* Patients with previously known allergies to the drugs to be used in the study,
* Infection near the puncture site,
* Patients with previous symptoms of neurological disease (TIA, syncope, dementia, etc.)
* Known coagulation disorders,
* Alcohol and drug use,
* Disorder of consciousness,
* Opioid use equal to or greater than 60 mg oral morphine equivalent per day,
* Patients with pre-existing neuropathic pain,
* Liver failure, renal failure, cardiac failure
* Morbid obesity (body mass index [BMI] > 35 kg m-2)
* Uncontrolled diabetes mellitus
* Women during pregnancy or breastfeeding
* Not approving the informed consent form

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery-15 (QoR-15) score | at the end of 24 hours postoperatively
  Quality of recovery-15 (QoR-15) score at 24 hours after surgery

SECONDARY OUTCOMES:
Postoperative opioid consumption | up to the first 24 hours postoperatively
  Total amount of morphine consumption during the first 24 hours after surgery. Patient controlled analgesia to be inserted.
Pain intensity score | 0, 2, 6, 12, 24 hours postoperatively.
  Postoperative pain assessed with verbal rating scale (VRS 0: no pain 10:pain as bad as can be ) at 0, 2, 6, 12, 24 hours postoperatively.
Postoperative nausea and vomiting | up to the first 24 hours postoperatively
  Nausea and vomiting intensity score measured by numeric rank score (0:no nausea and no vomiting, 1: have nausea, no vomiting, 2: once vomiting, 3: two or more vomiting).
Patient satisfaction | at the end of 24 hours postoperatively
  Patient satisfaction measured using a numeric rating scale 0 to 10 (0 = unsatisfied; 10 =very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Aylin Ceren Şanlı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided